CLINICAL TRIAL: NCT02408614
Title: Acute Effect of Exercise on Vascular Function
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401078
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Aging
MeSH Terms: interventions — High-Intensity Interval Training; Exercise Test

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Slow-paced walking: Subjects will complete 47 minutes of walking at slow pace.
  Interventions: Other: Slow-paced walking; Device: Treadmill
- Moderate-paced walking: Subjects will complete 47 minutes of walking at a moderate pace.
  Interventions: Other: Moderate-paced walking; Device: Treadmill
- Interval training: Subjects will complete 40 minutes of walking alternating between a moderate and fast pace.
  Interventions: Other: Interval Training; Device: Treadmill

INTERVENTIONS:
Other: Slow-paced walking — Subjects will complete 47 minutes of walking on a treadmill at a slow-pace.
  Groups: Slow-paced walking
Other: Moderate-paced walking — Subjects will complete 47 minutes of walking on a treadmill at a moderate pace.
  Groups: Moderate-paced walking
Other: Interval Training — Subjects will complete 40 minutes of walking on the treadmill alternating between a moderate and a fast pace.
  Groups: Interval training
Device: Treadmill

SUMMARY:
The study objectives are the following: 1) To examine the acute vascular responses to continuous low- and moderate-intensity exercise and interval training; and 2) To examine the influence of age and gender on these responses.

DETAILED DESCRIPTION:
The type, intensity and duration of exercise, fitness state, and timing of measurements have been reported to influence the acute vascular responses to exercise. However, little is known regarding the influence of interval training, aging and gender on these responses. The objectives of this study are: 1) to examine the acute vascular responses to continuous low- and moderate-intensity exercise and interval training; and 2) to examine the influence of age and gender on these responses. Subjects will perform the following 3 types of treadmill exercise in a random order: 1) slow-pace walking; 2) moderate-pace walking; and 3) interval training. Flow mediated dilation using high resolution ultrasonography and arterial stiffness using applanation tonometry will be measured before, immediately after and 1-hour after each acute bout of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 79 years of age
* Women will be premenopausal or postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years.
* Premenopausal women will be eumenorrheic.
* Able to give consent.

Exclusion Criteria:

* History of hepatic disease or infection with hepatitis B, C or HIV
* History of other relevant on-going or recurrent illness
* Recent (within 3 months) or recurrent hospitalizations
* Current intake of medications that may affect study results
* Use of tobacco products
* Premenopausal women taking oral contraceptives and postmenopausal women taking hormone replacement therapy.
* Pregnancy (positive urine pregnancy test) or lactation
* Perimenopausal women

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population including men and women 18 to 79 years of age
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function | Baseline, 15 minutes after exercise and 1 hour after exercise
  Brachial artery endothelium-dependent flow-mediated dilation to reactive hyperemia will be measured using high resolution ultrasonography. Brachial artery diameter and blood velocity will be measured before and after occluding the forearm for 5 minutes by inflating a cuff to 250 mmHg.

SECONDARY OUTCOMES:
Change in arterial stiffness | Baseline, 15 minutes after exercise and 1 hour after exercise
  Arterial stiffness (aortic pulse wave velocity and augmentation index) will be measured using applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovascular Physiology Laboratory, Gainesville, Florida, United States